CLINICAL TRIAL: NCT05278208
Title: Phase I/II Study of Lutathera in Patients With Recurrent and/or Progressive High-Grade Central Nervous System Tumors and Meningiomas That Demonstrate Uptake on DOTATATE PET
Brief Title: Lutathera for Treatment of Recurrent or Progressive High-Grade CNS Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT2007; FD-R-0532-01 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2022-02-07; First posted 2022-03-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: High Grade Glioma; Meningioma; Embryonal Tumor; Medulloblastoma; Anaplastic Ependymoma; Recurrent Diffuse Intrinsic Pontine Glioma; Recurrent Malignant Glioma; Recurrent Medulloblastoma; Recurrent Primary Central Nervous System Neoplasm; Refractory Diffuse Intrinsic Pontine Glioma; Refractory Malignant Glioma; Refractory Medulloblastoma; Refractory Primary Central Nervous System Neoplasm
Keywords: Somatostatin Receptor; DOTATATE; Lutathera
MeSH Terms: conditions — Glioma; Meningioma; Neoplasms, Germ Cell and Embryonal; Medulloblastoma; Ependymoma; Diffuse Intrinsic Pontine Glioma; Central Nervous System Neoplasms | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: Phase I (4 to <12 yrs) Lutathera (maximum dose of 200 mCi) once every 8 weeks (one cycle) for 4 cycles.
  Level 0: 150 mCi*(BSA/1.73m2). Level 1#: 200 mCi*(BSA/1.73m2). Level 2: 250 mCi*(BSA/1.73m2).
  #starting dose
  Phase II (12 to </=39 years) RP2D 200 mCi once every 8 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I-II (Experimental): Pediatric patients (4 to <12 years, Phase I) and adolescent and young adult patients (12 to </=39 years, Phase II) with recurrent/progressive high-grade central nervous system tumors and meningiomas that express SST2A and demonstrate uptake on DOTATATE PET will receive Lutathera once every 8 weeks (1 cycle) for a total of 4 doses over 8 months
  Phase I starting dose will be 200 mCi*(BSA/1.73m2), corresponding to the BSA-adjusted FDA approved adult Lutathera dosing. The first cycle will be used as the DLT period. Once MTD/RP2D is established, an efficacy expansion cohort of up to 10 patients will be opened to determine the preliminary efficacy of MTD/RP2D of Lutathera
  Phase II patients will receive the adult RP2D of 200 mCi every 8 weeks to determine the anti-tumor activity of Lutathera in this patient population, through evaluation of 6-month PFS as the primary efficacy endpoint. Response will be assessed on imaging (brain/spine MRI and DOTATATE PET) following every 1-2 cycles.
  Interventions: Drug: LUTATHERA® (Lutetium Lu 177 dotatate)

INTERVENTIONS:
Drug: LUTATHERA® (Lutetium Lu 177 dotatate) — Lutathera: IV administration maximum dose of 200 mCi once every 8 weeks (one cycle) for total of 4 cycles (8 months)
  Other Names: Lutathera

SUMMARY:
This study will evaluate the safety and efficacy of Lutathera (177Lu-DOTATATE) in patients with progressive or recurrent High-Grade Central Nervous System (CNS) tumors and meningiomas that demonstrate uptake on DOTATATE PET. The drug will be given intravenously once every 8 weeks for a total of up to 4 doses over 8 months in patients aged 4 to <12 years (Phase I) or 12 to </=39 years (Phase II) to test its safety and efficacy, respectively.

Funding Source - FDA OOPD (grant number FD-R-0532-01)

DETAILED DESCRIPTION:
Somatostatin receptors regulate cell growth through downstream modulation of both proliferation and apoptosis signaling pathways, and thus represent a potential therapeutic target. Lutathera (Lutetium [Lu]177 Dotatate) is a radionuclide therapy which binds type-2A somatostatin receptors (SST2A) and has recently gained FDA approval for the treatment of adult gastroenteropancreatic neuroendocrine tumors expressing SST2A.

High SST2A expression has been consistently observed in medulloblastoma and other embryonal tumors (75-100% of cases) as well as in some HGGs and anaplastic ependymomas (13-80%), with corresponding uptake on radiolabeled somatostatin receptor nuclear imaging (e.g. DOTATATE PET).

Emerging data has demonstrated treatment response (disease stabilization or regression) to somatostatin receptor-targeted therapy in children and young adults with relapsed medulloblastoma, HGG, meningioma, and brain metastases of neuroendocrine tumors, suggesting sufficient CNS penetration to achieve therapeutic benefit.

The proposed Phase I-II study will investigate the safety and efficacy of Lutathera treatment in patients whose tumors demonstrate uptake on DOTATATE PET (functional evidence of SST2A expression). In both Phase cohorts, Lutathera will be administered as an intravenous infusion on day 1 of each 8-week cycle for up to 4 cycles.

Phase I: (4 to <12 years) To determine the safety, define the dose-limiting toxicities, and establish the maximally tolerated dose (MTD)/ recommended Phase II dose (RP2D) of Lutathera in this patient population. The first cycle (first 8 weeks) will be used as the dose-limiting toxicity (DLT) observation period. The starting dose will be dose level 1, 200 mCi*(body surface area [BSA]/1.73m2), which corresponds to the BSA-adjusted FDA approved adult dosing of Lutathera (200 mCi every 8 weeks). Once the MTD/RP2D is established, an efficacy expansion cohort of up to 10 patients will be opened to determine the preliminary efficacy of the MTD/RP2D of Lutathera in this cohort.

Phase II: (12 to </=39 years) Enroll patients at the recommended adult dose of 200 mCi every 8 weeks to determine the anti-tumor activity of Lutathera at this dosing in this population. Response will be assessed on imaging (brain and/or spine MRI and DOTATATE PET) following every cycle or every other cycle.

ELIGIBILITY:
All participants must meet the following inclusion and exclusion criteria. No exceptions will be given. Imaging studies to establish eligibility must be done within three weeks prior to enrollment. All other clinical evaluations to establish eligibility (except for [68Ga]Ga-DOTATATE PET) must be done within 7 days prior to enrollment.

1. Screening Criteria

   1.1 Diagnosis Patient must have a diagnosis of primary high-grade CNS tumor (any histopathologic diagnosis that is WHO grade III-IV) or meningioma (any histologic grade) that is recurrent, progressive, or refractory. Note that patients with DIPG (based on radiographic/clinical diagnosis) who have undergone biopsy will be eligible with histologic diagnosis of grade II-IV infiltrating glioma. All tumors must have histologic verification either at the time of diagnosis or recurrence, except for patients meningioma who have not previously undergone biopsy or resection.

   Note: Refractory disease is defined as the presence of persistent abnormality on conventional MRI that is further distinguished by histology (biopsy or sample of lesion) or advanced imaging, OR as determined by the treating physician and discussed with the primary investigator prior to enrollment.

   1.2 Prior Therapy Patients must have recurred/progressed following prior standard therapy for their tumor. Note: Patients with meningioma, atypical meningioma, or anaplastic meningioma must have received at least surgical resection or radiation.

   1.3 Screening Consent Participant/legal guardian is willing to sign a screening consent for [68Ga]Ga-DOTATATE PET imaging. The screening consent is to be obtained according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.
2. Eligibility Criteria

   * Phase I Age Patient must be ≥ 4 and <12 years of age at the time of enrollment. Disease Status: Patients who participate in the efficacy expansion cohort must have bi-dimensionally measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions Patients with measurable extraneural disease only are also eligible.
   * Phase II Age Patient must be 12 to </=39 years at the time of enrollment.
3. Inclusion Criteria

   3.1 Uptake on [68Ga]Ga-DOTATATE PET Patients must have uptake on DOTATATE PET/CT in at least one tumor lesion (corresponding to known disease) equivalent to a Krenning score ≥2 (confirmed by central radiology review).

   3.2 Prior Therapy Patients must have recovered from the acute treatment related toxicities (defined as ≤ grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy, radiotherapy, or any other treatment modality prior to entering this study.

   3.3 Chemotherapy Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea.

   3.4 Investigational/Biologic Agent

   ●Biologic or investigational agent (anti-neoplastic): Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment.

   For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.

   ●Monoclonal Antibodies and agents with known prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.

   3.5 Radiation

   Patients must have had their last fraction of:
   * Craniospinal irradiation or total body irradiation or radiation to > 50% of pelvis > 3 months prior to enrollment.
   * Focal irradiation > 4 weeks prior to enrollment

   3.6 Stem Cell Transplant

   Patient must be:
   * ≥ 6 months since allogeneic stem cell transplant prior to enrollment with no evidence of active graft vs. host disease
   * ≥ 3 months since autologous stem cell transplant prior to enrollment

   3.7 Growth Factors Patients must be off all colony-forming growth factor(s) for at least 1 week prior to enrollment (e.g. filgrastim, sargramostim or erythropoietin). Two weeks must have elapsed if patients received long-acting formulations.

   3.8 Somatostatin analogs Patients must be off long-acting somatostatin analogs for at least 4 weeks and off short-acting somastatin analogs (i.e., octreotide) for at least 24 hours.

   3.9 Neurologic Status
   * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment, documented by a detailed neurological exam.
   * Patients with seizure disorders may be enrolled if seizures are well controlled.

   3.10 Performance Status Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within two weeks of enrollment must be ≥ 50. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score

   3.11 Organ Function

   Patients must have adequate organ and marrow function, both for eligibility for enrollment, and to begin each subsequent cycle of Lutathera, as defined below:
   * Adequate Bone Marrow Function as defined as:

     * Absolute neutrophil count ≥ 1.0 x 109 cells/ L
     * Platelets ≥100 x 109 cells/ L (unsupported, defined as no platelet transfusion within 7 days)
     * Hemoglobin ≥8 g/dl (may receive transfusions)
   * Adequate Renal Function as defined as:

     * Creatinine clearance or radioisotope GFR >70mL/min/1.73m2 OR
     * A serum creatinine based on (Schwartz et al. J. Peds, 106:522, 1985) age/gender as follows:

       1 to < 2 years: maximum serum creatinine 0.6 mg/dL for males and females. 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for males and females. 6 to < 10 years: maximum serum creatinine 1.0 mg/dL for males and females. 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for males and females. 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for males and 1.4 mg/dL for females.

       ≥ 16 years: maximum serum creatinine 1.7 mg/dL for males and 1.4 mg/dL for females.
   * Adequate Liver Function as defined as:

     * Total bilirubin ≤ 3 times institutional upper limit of normal (ULN) for age
     * AST(SGOT)/ALT(SGPT) ≤ 3 times institutional ULN
     * Serum albumin ≥ 2g/dL
     * Coagulation parameters: INR <1.5 times ULN and aPTT <1.5 times ULN unless patients are receiving therapeutic anticoagulation which affects these parameters
   * Adequate Cardiac Function as defined as:

     * Ejection fraction of ≥ 55% by echocardiogram
     * Serum electrolytes (Sodium, Potassium, Chloride) within institutional limits of normal (patients can be on enteral supplementation)

   3.12 Corticosteroids Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment, with a maximum dexamethasone dose of 2.5mg/m2/day.

   3.13 Pregnancy Status Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   3.14 Pregnancy Prevention Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for at least 7 months after drug cessation in females of childbearing potential and for at least 4 months after drug cessation in males of child fathering potential.

   3.15 Informed Consent The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.
4. Exclusion Criteria

   4.1 Confirmed bone marrow metastatic disease Patients with confirmed metastatic disease to bone marrow are ineligible.

   4.2 Presence of bulky disease Patients with bulky disease on imaging as described below are ineligible. Treating physicians are encouraged to request a rapid central imaging review to confirm fulfillment of these criteria if there are questions or concerns.

   Bulky disease is defined as:
   * Tumor with evidence of clinically significant uncal herniation or midline shift.
   * Tumor with diameter of >5cm in one dimension on T2/FLAIR.
   * Tumor that in the opinion of the site investigator shows significant mass effect in either the brain or spine.

   Note that patients with metastatic or multi-focal disease (with exception of bone marrow) are eligible as long as no sites of disease meet above criteria for bulky disease.

   4.3 Breast-feeding Nursing mothers are excluded from this study. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Lutathera.

   4.4 Concurrent Illness
   * Patients with a history of any other malignancy, except patients with a secondary brain tumor if the patient's prior malignancy has been in remission for at least 5 years from the end of treatment.
   * Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
   * Patients with type I diabetes.

   4.5 Concomitant Medications
   * Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible.
   * Prior or current treatment with 177Lu-DOTATATE/TOC or 90Y-DOTATATE/TOC.

   4.6 Prisoners will be excluded from this study.

   4.7 Inability to participate: Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits, obtain follow-up studies required to assess toxicity to therapy, or adhere to drug administration plan, other study procedures, and study restrictions.
5. Inclusion of Women and Minorities Both males and females of all races and ethnic groups are eligible for this study.

Ages: 4 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Estimate MTD of Lutathera in pediatric CNS patients 4 to <12 years | up to 8 months
  To estimate the maximum tolerated dose (MTD) of Lutathera in pediatric patients between 4 and 12 to </=39 yearsof age with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET.
Estimate RP2D of Lutathera in pediatric CNS patients 4 to <12 years | up to 8 months
  To estimate the recommended Phase II dose (RP2D) of Lutathera in pediatric patients between 4 and 12 to </=39 years of age with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET.
Calculate the incidence of treatment related adverse events as assessed by CTCAE v5.0 in pediatric (4 to <12 yo) CNS patients treated with Lutathera | up to 2 months
  To define and describe the toxicities of Lutathera in pediatric patients with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET. This will include calculating the number of participants with Lutathera-related adverse events as assessed by CTCAE v 5.0
Assess PFS of Lutathera in CNS patients 12 to </=39 years | up to 6 months
  To assess efficacy, evaluated by 6 month progression-free survival, of treatment with Lutathera in adolescent and young adult patients age 12 to </=39 years with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET

SECONDARY OUTCOMES:
Objective Response Rate of Lutathera in CNS patients 12 to </=39 years | up to 8 months
  To evaluate the objective response rate of Lutathera in adolescent and young adult patients age 12 to </=39 years with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET.
Calculate the incidence of treatment related adverse events as assessed by CTCAE v5.0 in CNS patients 12 </=39 years treated with Lutathera | up to 8 months
  To establish the safety and toxicity of Lutathera 200 mCi every 8-week dosing in adolescent and young adult patients age 12 to </=39 years with recurrent and/or progressive high-grade CNS tumors or meningiomas that demonstrate uptake on DOTATATE PET. This will include calculating the number of participants with, as well as severity and frequency of, Lutathera-related adverse events as assessed by CTCAE v 5.0

OTHER OUTCOMES:
Anti-tumor activity of Lutathera | up to 8 months
  Document anti-tumor activity of Lutathera through assessment of ORR, PFS in patients with recurrent or progressive High-Grade CNS tumors or meningiomas
Prevalence of SST2A expression in patients with different high-grade CNS tumors | up to 8 months
  Describe prevalence and heterogeneity of SST2A expression (IHC) in patients with recurrent or progressive High-Grade CNS tumors or meningiomas
Correlation of SST2A expression with clinical and molecular features in high-grade CNS tumor patients treated with Lutathera | up to 8 months
  Assess correlation of SST2A expression with uptake on DOTATATE PET, response to Lutathera therapy, and relevant clinical and molecular features within the confines of a Phase I/II study in patients with recurrent or progressive High-Grade CNS tumors or meningiomas treated with Lutathera

CONTACTS AND LOCATIONS:
Overall Officials: Margot Lazow, MD, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotteveel JJ, Colon EJ. Preliminary note: vertebral-Doppler sonography in near sudden infant death syndrome (NSIDS). Pediatr Radiol. 1985;15(2):95-7. doi: 10.1007/BF02388711. PMID 3883302
- [Background] Theodoropoulou M, Stalla GK. Somatostatin receptors: from signaling to clinical practice. Front Neuroendocrinol. 2013 Aug;34(3):228-52. doi: 10.1016/j.yfrne.2013.07.005. Epub 2013 Jul 18. PMID 23872332
- [Background] Khera DC, Herschman BR, Sosa F. Tetracycline-induced esophageal ulcers. Report of two cases. Postgrad Med. 1980 Oct;68(4):113, 115. doi: 10.1080/00325481.1980.11715564. PMID 6448409
- [Background] Reubi JC, Schar JC, Waser B, Wenger S, Heppeler A, Schmitt JS, Macke HR. Affinity profiles for human somatostatin receptor subtypes SST1-SST5 of somatostatin radiotracers selected for scintigraphic and radiotherapeutic use. Eur J Nucl Med. 2000 Mar;27(3):273-82. doi: 10.1007/s002590050034. PMID 10774879
- [Background] Vaidyanathan G, Affleck DJ, Zhao XG, Keir ST, Zalutsky MR. [Lu]-DOTA-Tyr-octreotate: A Potential Targeted Radiotherapeutic for the Treatment of Medulloblastoma. Curr Radiopharm. 2010;3(1):29-36. doi: 10.2174/1874471011003010029. PMID 21243098
- [Background] Hauser P, Hanzely Z, Mathe D, Szabo E, Barna G, Sebestyen A, Jeney A, Schuler D, Fekete G, Garami M. Effect of somatostatin analogue octreotide in medulloblastoma in xenograft and cell culture study. Pediatr Hematol Oncol. 2009 Jul-Aug;26(5):363-74. doi: 10.1080/08880010902973293. PMID 19579083
- [Background] Pinski J, Schally AV, Halmos G, Szepeshazi K, Groot K. Somatostatin analogues and bombesin/gastrin-releasing peptide antagonist RC-3095 inhibit the growth of human glioblastomas in vitro and in vivo. Cancer Res. 1994 Nov 15;54(22):5895-901. PMID 7954420
- [Background] Volante M, Brizzi MP, Faggiano A, La Rosa S, Rapa I, Ferrero A, Mansueto G, Righi L, Garancini S, Capella C, De Rosa G, Dogliotti L, Colao A, Papotti M. Somatostatin receptor type 2A immunohistochemistry in neuroendocrine tumors: a proposal of scoring system correlated with somatostatin receptor scintigraphy. Mod Pathol. 2007 Nov;20(11):1172-82. doi: 10.1038/modpathol.3800954. Epub 2007 Sep 14. PMID 17873898
- [Background] Fruhwald MC, O'Dorisio MS, Pietsch T, Reubi JC. High expression of somatostatin receptor subtype 2 (sst2) in medulloblastoma: implications for diagnosis and therapy. Pediatr Res. 1999 May;45(5 Pt 1):697-708. doi: 10.1203/00006450-199905010-00016. PMID 10231868
- [Background] Remke M, Hering E, Gerber NU, Kool M, Sturm D, Rickert CH, Gerss J, Schulz S, Hielscher T, Hasselblatt M, Jeibmann A, Hans V, Ramaswamy V, Taylor MD, Pietsch T, Rutkowski S, Korshunov A, Monoranu CM, Fruhwald MC. Somatostatin receptor subtype 2 (sst(2)) is a potential prognostic marker and a therapeutic target in medulloblastoma. Childs Nerv Syst. 2013 Aug;29(8):1253-62. doi: 10.1007/s00381-013-2142-4. Epub 2013 May 16. PMID 23677175
- [Background] Guyotat J, Champier J, Pierre GS, Jouvet A, Bret P, Brisson C, Belin MF, Signorelli F, Montange MF. Differential expression of somatostatin receptors in medulloblastoma. J Neurooncol. 2001 Jan;51(2):93-103. doi: 10.1023/a:1010624702443. PMID 11386415
- [Background] Johnson MD, O'Connell MJ, Silberstein H, Korones D. Differential expression of somatostatin receptors, P44/42 MAPK, and mTOR activation in medulloblastomas and primitive neuroectodermal tumors. Appl Immunohistochem Mol Morphol. 2013 Dec;21(6):532-8. doi: 10.1097/PAI.0b013e3182813724. PMID 23455179
- [Background] Muller HL, Fruhwald MC, Scheubeck M, Rendl J, Warmuth-Metz M, Sorensen N, Kuhl J, Reubi JC. A possible role for somatostatin receptor scintigraphy in the diagnosis and follow-up of children with medulloblastoma. J Neurooncol. 1998 May;38(1):27-40. doi: 10.1023/a:1005961302340. PMID 9540055
- [Background] Fruhwald MC, Rickert CH, O'Dorisio MS, Madsen M, Warmuth-Metz M, Khanna G, Paulus W, Kuhl J, Jurgens H, Schneider P, Muller HL. Somatostatin receptor subtype 2 is expressed by supratentorial primitive neuroectodermal tumors of childhood and can be targeted for somatostatin receptor imaging. Clin Cancer Res. 2004 May 1;10(9):2997-3006. doi: 10.1158/1078-0432.ccr-03-0083. PMID 15131035
- [Background] Feindt J, Becker I, Blomer U, Hugo HH, Mehdorn HM, Krisch B, Mentlein R. Expression of somatostatin receptor subtypes in cultured astrocytes and gliomas. J Neurochem. 1995 Nov;65(5):1997-2005. doi: 10.1046/j.1471-4159.1995.65051997.x. PMID 7595483
- [Background] Held-Feindt J, Krisch B, Mentlein R. Molecular analysis of the somatostatin receptor subtype 2 in human glioma cells. Brain Res Mol Brain Res. 1999 Jan 22;64(1):101-7. doi: 10.1016/s0169-328x(98)00312-x. PMID 9889335
- [Background] Kiviniemi A, Gardberg M, Kivinen K, Posti JP, Vuorinen V, Sipila J, Rahi M, Sankinen M, Minn H. Somatostatin receptor 2A in gliomas: Association with oligodendrogliomas and favourable outcome. Oncotarget. 2017 Jul 25;8(30):49123-49132. doi: 10.18632/oncotarget.17097. PMID 28467778
- [Background] Appay R, Tabouret E, Touat M, Carpentier C, Colin C, Ducray F, Idbaih A, Mokhtari K, Uro-Coste E, Dehais C, Figarella-Branger D; POLA network. Somatostatin receptor 2A protein expression characterizes anaplastic oligodendrogliomas with favorable outcome. Acta Neuropathol Commun. 2018 Sep 7;6(1):89. doi: 10.1186/s40478-018-0594-1. PMID 30193580
- [Background] Cervera P, Videau C, Viollet C, Petrucci C, Lacombe J, Winsky-Sommerer R, Csaba Z, Helboe L, Daumas-Duport C, Reubi JC, Epelbaum J. Comparison of somatostatin receptor expression in human gliomas and medulloblastomas. J Neuroendocrinol. 2002 Jun;14(6):458-71. doi: 10.1046/j.1365-2826.2002.00801.x. PMID 12047721
- [Background] Lapa C, Linsenmann T, Luckerath K, Samnick S, Herrmann K, Stoffer C, Ernestus RI, Buck AK, Lohr M, Monoranu CM. Tumor-associated macrophages in glioblastoma multiforme-a suitable target for somatostatin receptor-based imaging and therapy? PLoS One. 2015 Mar 25;10(3):e0122269. doi: 10.1371/journal.pone.0122269. eCollection 2015. PMID 25807228
- [Background] Schulz S, Pauli SU, Schulz S, Handel M, Dietzmann K, Firsching R, Hollt V. Immunohistochemical determination of five somatostatin receptors in meningioma reveals frequent overexpression of somatostatin receptor subtype sst2A. Clin Cancer Res. 2000 May;6(5):1865-74. PMID 10815909
- [Background] Savelli G, Muni A. Somatostatin Receptors in an Anaplastic Oligodendroglioma Relapse Evidenced By 68Ga DOTANOC PET/CT. Clin Nucl Med. 2015 Jul;40(7):e363-5. doi: 10.1097/RLU.0000000000000816. PMID 26018682
- [Background] Collamati F, Pepe A, Bellini F, Bocci V, Chiodi G, Cremonesi M, De Lucia E, Ferrari ME, Frallicciardi PM, Grana CM, Marafini M, Mattei I, Morganti S, Patera V, Piersanti L, Recchia L, Russomando A, Sarti A, Sciubba A, Senzacqua M, Solfaroli Camillocci E, Voena C, Pinci D, Faccini R. Toward radioguided surgery with beta- decays: uptake of a somatostatin analogue, DOTATOC, in meningioma and high-grade glioma. J Nucl Med. 2015 Jan;56(1):3-8. doi: 10.2967/jnumed.114.145995. Epub 2014 Dec 11. PMID 25500828
- [Background] Khanna G, O'Dorisio MS, Menda Y, Glasier C, Deyoung B, Smith BJ, Graham M, Juweid M. Somatostatin receptor scintigraphy in surveillance of pediatric brain malignancies. Pediatr Blood Cancer. 2008 Mar;50(3):561-6. doi: 10.1002/pbc.21194. PMID 17387742
- [Background] Marincek N, Radojewski P, Dumont RA, Brunner P, Muller-Brand J, Maecke HR, Briel M, Walter MA. Somatostatin receptor-targeted radiopeptide therapy with 90Y-DOTATOC and 177Lu-DOTATOC in progressive meningioma: long-term results of a phase II clinical trial. J Nucl Med. 2015 Feb;56(2):171-6. doi: 10.2967/jnumed.114.147256. Epub 2015 Jan 15. PMID 25593116
- [Background] de Jong M, Breeman WA, Bernard BF, Bakker WH, Schaar M, van Gameren A, Bugaj JE, Erion J, Schmidt M, Srinivasan A, Krenning EP. [177Lu-DOTA(0),Tyr3] octreotate for somatostatin receptor-targeted radionuclide therapy. Int J Cancer. 2001 Jun 1;92(5):628-33. doi: 10.1002/1097-0215(20010601)92:53.0.co;2-l. PMID 11340564
- [Background] Galvis L, Gonzalez D, Bonilla C. Relapsed High-Risk Medulloblastoma: Stable Disease after Two Years of Treatment with Somatostatin Analog - Case Report. Cureus. 2016 Jan 4;8(1):e446. doi: 10.7759/cureus.446. PMID 26918214
- [Background] Glas M, Hennemann B, Hirschmann B, Marienhagen J, Schmidt-Wolf I, Herrlinger U, Bogdahn U, Hau P. Complete response after treatment with a somatostatin analogue in an adult patient with recurrent medulloblastoma. Acta Oncol. 2008;47(3):479-80. doi: 10.1080/02841860701678795. Epub 2007 Oct 12. No abstract available. PMID 17934891
- [Background] Florio T. Molecular mechanisms of the antiproliferative activity of somatostatin receptors (SSTRs) in neuroendocrine tumors. Front Biosci. 2008 Jan 1;13:822-40. doi: 10.2741/2722. PMID 17981589
- [Background] Menda Y, O'Dorisio MS, Kao S, Khanna G, Michael S, Connolly M, Babich J, O'Dorisio T, Bushnell D, Madsen M. Phase I trial of 90Y-DOTATOC therapy in children and young adults with refractory solid tumors that express somatostatin receptors. J Nucl Med. 2010 Oct;51(10):1524-31. doi: 10.2967/jnumed.110.075226. Epub 2010 Sep 16. PMID 20847174
- [Background] Dutour A, Kumar U, Panetta R, Ouafik L, Fina F, Sasi R, Patel YC. Expression of somatostatin receptor subtypes in human brain tumors. Int J Cancer. 1998 May 29;76(5):620-7. doi: 10.1002/(sici)1097-0215(19980529)76:53.0.co;2-s. PMID 9610716
- [Background] Hosono M, Ikebuchi H, Nakamura Y, Nakamura N, Yamada T, Yanagida S, Kitaoka A, Kojima K, Sugano H, Kinuya S, Inoue T, Hatazawa J. Manual on the proper use of lutetium-177-labeled somatostatin analogue (Lu-177-DOTA-TATE) injectable in radionuclide therapy (2nd ed.). Ann Nucl Med. 2018 Apr;32(3):217-235. doi: 10.1007/s12149-018-1230-7. Epub 2018 Jan 15. PMID 29333565
- [Background] Hamiditabar M, Ali M, Roys J, Wolin EM, O'Dorisio TM, Ranganathan D, Tworowska I, Strosberg JR, Delpassand ES. Peptide Receptor Radionuclide Therapy With 177Lu-Octreotate in Patients With Somatostatin Receptor Expressing Neuroendocrine Tumors: Six Years' Assessment. Clin Nucl Med. 2017 Jun;42(6):436-443. doi: 10.1097/RLU.0000000000001629. PMID 28263217
- [Background] John M, Meyerhof W, Richter D, Waser B, Schaer JC, Scherubl H, Boese-Landgraf J, Neuhaus P, Ziske C, Molling K, Riecken EO, Reubi JC, Wiedenmann B. Positive somatostatin receptor scintigraphy correlates with the presence of somatostatin receptor subtype 2. Gut. 1996 Jan;38(1):33-9. doi: 10.1136/gut.38.1.33. PMID 8566856
- [Background] Diakatou E, Alexandraki KI, Tsolakis AV, Kontogeorgos G, Chatzellis E, Leonti A, Kaltsas GA. Somatostatin and dopamine receptor expression in neuroendocrine neoplasms: correlation of immunohistochemical findings with somatostatin receptor scintigraphy visual scores. Clin Endocrinol (Oxf). 2015 Sep;83(3):420-8. doi: 10.1111/cen.12775. Epub 2015 Apr 24. PMID 25808161
- [Background] Miederer M, Seidl S, Buck A, Scheidhauer K, Wester HJ, Schwaiger M, Perren A. Correlation of immunohistopathological expression of somatostatin receptor 2 with standardised uptake values in 68Ga-DOTATOC PET/CT. Eur J Nucl Med Mol Imaging. 2009 Jan;36(1):48-52. doi: 10.1007/s00259-008-0944-5. Epub 2008 Sep 20. PMID 18807033
- [Background] Korner M, Waser B, Schonbrunn A, Perren A, Reubi JC. Somatostatin receptor subtype 2A immunohistochemistry using a new monoclonal antibody selects tumors suitable for in vivo somatostatin receptor targeting. Am J Surg Pathol. 2012 Feb;36(2):242-52. doi: 10.1097/PAS.0b013e31823d07f3. PMID 22251942
- [Background] Qian ZR, Li T, Ter-Minassian M, Yang J, Chan JA, Brais LK, Masugi Y, Thiaglingam A, Brooks N, Nishihara R, Bonnemarie M, Masuda A, Inamura K, Kim SA, Mima K, Sukawa Y, Dou R, Lin X, Christiani DC, Schmidlin F, Fuchs CS, Mahmood U, Ogino S, Kulke MH. Association Between Somatostatin Receptor Expression and Clinical Outcomes in Neuroendocrine Tumors. Pancreas. 2016 Nov;45(10):1386-1393. doi: 10.1097/MPA.0000000000000700. PMID 27622342
- [Background] Reubi JC, Laissue JA, Waser B, Steffen DL, Hipkin RW, Schonbrunn A. Immunohistochemical detection of somatostatin sst2a receptors in the lymphatic, smooth muscular, and peripheral nervous systems of the human gastrointestinal tract: facts and artifacts. J Clin Endocrinol Metab. 1999 Aug;84(8):2942-50. doi: 10.1210/jcem.84.8.5878. PMID 10443702
- [Background] Mehta S, de Reuver PR, Gill P, Andrici J, D'Urso L, Mittal A, Pavlakis N, Clarke S, Samra JS, Gill AJ. Somatostatin Receptor SSTR-2a Expression Is a Stronger Predictor for Survival Than Ki-67 in Pancreatic Neuroendocrine Tumors. Medicine (Baltimore). 2015 Oct;94(40):e1281. doi: 10.1097/MD.0000000000001281. PMID 26447992
- [Background] Okuwaki K, Kida M, Mikami T, Yamauchi H, Imaizumi H, Miyazawa S, Iwai T, Takezawa M, Saegusa M, Watanabe M, Koizumi W. Clinicopathologic characteristics of pancreatic neuroendocrine tumors and relation of somatostatin receptor type 2A to outcomes. Cancer. 2013 Dec 1;119(23):4094-102. doi: 10.1002/cncr.28341. Epub 2013 Sep 10. PMID 24022344
- [Background] Corleto VD, Falconi M, Panzuto F, Milione M, De Luca O, Perri P, Cannizzaro R, Bordi C, Pederzoli P, Scarpa A, Delle Fave G. Somatostatin receptor subtypes 2 and 5 are associated with better survival in well-differentiated endocrine carcinomas. Neuroendocrinology. 2009;89(2):223-30. doi: 10.1159/000167796. Epub 2008 Oct 31. PMID 18974627
- [Background] Moertel CL, Reubi JC, Scheithauer BS, Schaid DJ, Kvols LK. Expression of somatostatin receptors in childhood neuroblastoma. Am J Clin Pathol. 1994 Dec;102(6):752-6. doi: 10.1093/ajcp/102.6.752. PMID 7801887
- [Background] Haug AR, Auernhammer CJ, Wangler B, Schmidt GP, Uebleis C, Goke B, Cumming P, Bartenstein P, Tiling R, Hacker M. 68Ga-DOTATATE PET/CT for the early prediction of response to somatostatin receptor-mediated radionuclide therapy in patients with well-differentiated neuroendocrine tumors. J Nucl Med. 2010 Sep;51(9):1349-56. doi: 10.2967/jnumed.110.075002. Epub 2010 Aug 18. PMID 20720050
- [Background] Kwekkeboom DJ, Krenning EP. Somatostatin receptor imaging. Semin Nucl Med. 2002 Apr;32(2):84-91. doi: 10.1053/snuc.2002.31022. PMID 11965603
- [Background] Kwekkeboom DJ, Teunissen JJ, Bakker WH, Kooij PP, de Herder WW, Feelders RA, van Eijck CH, Esser JP, Kam BL, Krenning EP. Radiolabeled somatostatin analog [177Lu-DOTA0,Tyr3]octreotate in patients with endocrine gastroenteropancreatic tumors. J Clin Oncol. 2005 Apr 20;23(12):2754-62. doi: 10.1200/JCO.2005.08.066. PMID 15837990
- [Background] Hofman MS, Lau WF, Hicks RJ. Somatostatin receptor imaging with 68Ga DOTATATE PET/CT: clinical utility, normal patterns, pearls, and pitfalls in interpretation. Radiographics. 2015 Mar-Apr;35(2):500-16. doi: 10.1148/rg.352140164. PMID 25763733